CLINICAL TRIAL: NCT00180505
Title: Non-Randomized, Prospective, Multi-center Evaluation of the ABSOLUTE™ .035 Peripheral Self-Expanding Stent System for Occluded or Stenotic Superficial Femoral or Proximal Popliteal Arteries
Brief Title: ASSESS Study: Evaluation of ABSOLUTE™ Stent System for Occluded Arteries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Ellen Travis, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-100
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Peripheral Vascular Diseases
Keywords: Peripheral Artery Disease; Restenosis Rate; Patency Rates; Self-Expandable Nitinol Stents; Stent Fractures
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): The purpose of the ASSESS Registry is to investigate the performance of the ABSOLUTE™ .035 Peripheral Self-Expanding Stent System (ABSOLUTE™ Stent) in preventing restenosis of occluded or stenotic superficial femoral or proximal popliteal arteries.
  Interventions: Device: ABSOLUTE™: Self-Expandable Peripheral Nitinol Stent

INTERVENTIONS:
Device: ABSOLUTE™: Self-Expandable Peripheral Nitinol Stent — A prospective, non-randomized, multi-center study to investigate the performance of the ABSOLUTE™ .035 Peripheral Self-Expanding Stent System (ABSOLUTE™ Stent) in preventing restenosis of occluded or stenotic superficial femoral or proximal popliteal arteries. Follow up at 30, 180, 270, 365 days and 2 years.

SUMMARY:
The purpose of this study is to investigate the performance of the ABSOLUTE™ .035 peripheral self-expanding stent system in preventing restenosis of occluded or stenotic superficial femoral or proximal popliteal arteries.

DETAILED DESCRIPTION:
The treatment of stenosis in superficial femoral arteries and/or proximal popliteal arteries with stenting is associated with high restenosis rates, especially with the first generation stents (stainless steel). Currently, self-expandable nitinol stents are commercialized which lead to higher primary patency rates as compared to the first generation stents, even in longer lesions. However, until now most data available are retrospective and uni-center. The ASSESS study is a prospective multi-center study investigating the performance (restenosis rate, patency rates) of the ABSOLUTE™. 035 peripheral self-expandable stent in longer lesions (lesion length from 4.00 mm to 200.00 mm).

Moreover, literature shows stent fracture in nitinol stents, with a possible clinical relationship. For this reason, the ASSESS study will analyze the stent fractures of the ABSOLUTE™ stent, and a possible relationship between stent fracture and restenosis.

ELIGIBILITY:
Inclusion Criteria:

* De novo lesion of the superficial femoral artery (SFA) or proximal popliteal artery within the following parameters:

  * 10 mm distal to the origin of the profunda femoris (= 10 mm from the femoral bifurcation in the SFA) and
  * 20 mm from the proximal margin of the intercondylar fossa.
* Patients must have symptomatic leg ischemia, requiring treatment of the superficial femoral/proximal popliteal vessel
* Target vessel reference diameter visually estimated to be > 4.0 mm and < 7.0 mm
* Target lesion length visually estimated to be > 40 mm and < 200 mm
* If the patient has a contralateral SFA or contralateral proximal popliteal lesion, this lesion can be treated as a non-target lesion. The time and way of treatment of the non-target lesion will be left up to the discretion of the investigator
* At least one-vessel run-off to the foot confirmed by baseline angiography
* Patent common iliac artery, common femoral artery and profunda confirmed by baseline angiography. The patent common iliac artery can be obtained during the index procedure by a successful treatment prior to the treatment of the target lesion. Successful treatment being defined as attainment of final residual diameter stenosis of < 30% without death, stroke, bleeding requiring > 2 units transfusion, or any other complication which was device or procedure related.
* Patient is acceptable candidate for femoral-popliteal artery bypass surgery

Exclusion Criteria:

* Previous ipsilateral femoro-popliteal or femoro-tibial surgery
* Presence of a stent in the target vessel
* Prescheduled staged procedures of multiple lesions within the ipsilateral iliac or ipsilateral popliteal arteries within 30 days after the index procedure
* Co-existing aneurysmal disease of the abdominal aorta or iliac or popliteal arteries
* Acute thrombophlebitis or deep vein thrombus
* Any immunosuppressive disorders, groin infection, or acute systemic infection due to any cause or any viral or bacterial infection
* Significant gastrointestinal (GI) bleed within the past month that would contraindicate the use of anti-platelet therapy
* Hemodynamic instability
* Target lesion is restenotic from previous intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Restenosis rate (diameter stenosis ≥ 50% as determined by Duplex ultrasound). | At 180 days

SECONDARY OUTCOMES:
Clinically driven target lesion revascularization | at 12 and 24 month follow-up
Target lesion primary, primary assisted and secondary patency rates | at 6, 12 and 24 month follow-up
Major complications | at 1, 6, 12 and 24 month follow-up
Angiographic binary restenosis rate in a subset of patients | at 9 month follow-up
Device and procedure success | Acute
Vascular and bleeding complications (local and puncture site) | 1, 6, 12, 24 months
Stent fracture determined by biplane X-ray | at 12 month follow-up
Restenosis rate at 365 days, and 2 years (diameter stenosis ≥ 50% as determined by Duplex ultrasound) | 365 days and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, M.D., Principal Investigator — Herzzentrum Bad Krozingen, Germany
Locations (13):
- Austria (2):
  - Landeskrankenhaus Klagenfurt, Klagenfurt
  - Allgemeines Krankenhaus der Stadt Wien (AKH Wien), Vienna
- CHR de Namur, Namur, Belgium
- France (2):
  - Polyclinique Louis Pasteur, Essey-lès-Nancy
  - Hôpital Pontchaillou- CHU, Rennes
- Germany (3):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - Universitäres Herz & Gefässzentrum Hamburg, Hamburg
  - Herzzentrum Leipzig, Leipzig
- Papageorgiou Hospital, Thessaloniki, Greece
- Italy (3):
  - Nuovo Ospedale Civile Sant' Agostino, Baggiovara (Modena)
  - Casa di Cura Montevergine, Mercogliano
  - Policlinico San Matteo, Pavia
- Hospital de Donostia, Donostia / San Sebastian, Spain